CLINICAL TRIAL: NCT00091130
Title: An Exploratory Study to Evaluate the Effect of HPV 16 Vaccine on the Reduction of Viral Load in HPV 16 Positive Women With Persistent Viral Infection, But Low Grade Disease (ASCUS/LSIL)
Brief Title: SGN-00101 Vaccine in Treating Human Papillomavirus in Patients Who Have Abnormal Cervical Cells
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2012-02623; UCI#02-55; N01CN25139 (Other Grant/Funding Number: US NIH Grant/Contract Award Number); CDR0000383786 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-09-07; First posted 2004-09-08 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-03

CONDITIONS: Atypical Squamous Cells of Undetermined Significance; Cervical Cancer; High-grade Squamous Intraepithelial Lesion; Low-grade Squamous Intraepithelial Lesion
MeSH Terms: conditions — Atypical Squamous Cells of the Cervix; Uterine Cervical Neoplasms; Squamous Intraepithelial Lesions

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (SGN-00101) (Experimental): Patients receive SGN-00101 vaccine SC on day 1 of weeks 1, 4, and 8 for a maximum of 3 injections in the absence of unacceptable toxicity or the development of an invasive malignancy or serious illness.
  Interventions: Biological: HspE7; Other: laboratory biomarker analysis
- Arm II (placebo) (Placebo Comparator): Patients receive placebo vaccine SC on day 1 of weeks 1, 4, and 8 for a maximum of 3 injections in the absence of unacceptable toxicity or the development of an invasive malignancy or serious illness.
  Interventions: Other: placebo; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: HspE7 — Given SC
  Other Names: HPV 16 E7/HSP65 Vaccine; HPV E7 Peptide Epitope Vaccine; SGN-00101
  Arms: Arm I (SGN-00101)
Other: placebo — Given SC
  Other Names: PLCB
  Arms: Arm II (placebo)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial is studying how well SGN-00101 vaccine works compared to a placebo in treating human papillomavirus and preventing cervical cancer in patients with abnormal cervical cells. Vaccines, such as SGN-00101, may make the body build an immune response to kill human papillomavirus and abnormal cervical cells and may be effective in preventing cervical cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the effectiveness of SGN-00101 vaccine vs placebo in reducing the human papillomavirus (HPV)-16 viral load in patients with atypical squamous cells of undetermined significance (ASCUS) or low-grade squamous intraepithelial lesions (LSIL) of the cervix with persistent HPV-16 infection who are at increased risk for developing a high-grade squamous intraepithelial lesion or invasive cervical cancer.

II. Compare the natural history of HPV-16 viral load in patients treated with these regimens.

III. Compare the effect of HPV-16 variants on viral load response in patients treated with these regimens.

IV. Compare the relative effectiveness of these regimens on the regression of cervical cellular atypias (based on Pap test results), in terms of the regression of cytologic findings of LSIL and ASCUS to normal findings and resolution or regression of colposcopically defined cervicovaginal lesions, in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive SGN-00101 vaccine subcutaneously (SC) on day 1 of weeks 1, 4, and 8 for a maximum of 3 injections in the absence of unacceptable toxicity or the development of an invasive malignancy or serious illness.

ARM II: Patients receive placebo vaccine SC on day 1 of weeks 1, 4, and 8 for a maximum of 3 injections in the absence of unacceptable toxicity or the development of an invasive malignancy or serious illness.

Patients are followed at 12, 24, and 52 weeks after the last vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for 1 of the following groups:

  * Prospective group, meeting the following criteria:

    * Evidence of atypical squamous cells of undetermined significance (ASCUS) or low-grade squamous intraepithelial lesions (LSIL) by Pap test
    * Human papillomavirus (HPV)-16-positive by polymerase chain reaction (PCR) and PGMY09/PGMY11 oligonucleotide primers viral load assay
  * Medical records-based group, meeting the following criteria:

    * Medical-record evidence of ASCUS or LSIL by Pap test within the past 6-12 months
    * Meets 1 of the following criteria:

      * Liquid-cytology findings of ASCUS or LSIL
      * Colposcopic evidence of a LSIL by the Reid Index score of 1-5
    * Historically persistent HPV-16-infection by PCR and HPV reverse transcription (RT)-PCR
    * No evidence of high-grade squamous intraepithelial lesions (HSIL) by colposcopy (Reid Index ≥ 6)
    * Reports no sex partner change since last index Pap screening test
  * Specimen-based group, meeting the following criteria:

    * Medical-record evidence of ASCUS or LSIL by Pap test within the past 6-12 months

      * Liquid-based cytology specimen available
    * Meets 1 of the following criteria:

      * Liquid-cytology findings of ASCUS or LSIL
      * Colposcopic evidence of a LSIL by the Reid Index score of 1-5
    * Historically persistent HPV-16-infection by PCR and, where measurable, HPV RT-PCR showing no greater than 3-fold reduction over the index liquid-cytology specimen
    * No evidence of HSIL by colposcopy (Reid Index ≥ 6)
* Menstrual period occurred at least once within the past 52 weeks
* No HSIL by Pap test within the past year
* Performance status - ECOG 0
* No severe or unstable coagulation
* Hepatitis B surface antigen negative
* Hepatitis C antibody negative
* No angina
* No heart failure
* No other cardiac condition
* No respiratory condition
* No asthma
* No immunological disorders (e.g., lupus, diabetes, multiple sclerosis, or myasthenia gravis)
* Not immunocompromised, suggestive of severe immune deficiency
* HIV negative
* No AIDS
* No active infection, defined as fever > 100° F
* No syphilis
* No severe allergic reactions (anaphylactic response) to drugs or any other allergen
* No history of allergy to any vaccine constituents, including cell- or tissue-system elements used to prepare the vaccine (e.g., bread products, yeast, or recombinant DNA technology using yeast systems)
* Must agree to use effective form of contraception throughout vaccination period
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during vaccination period and for 5 months after study treatment
* No sexual intercourse within 48 hours of virus specimen collection during study visits
* No objects (e.g., tampons, douche, suppositories, fingers, or toes) within the vagina or rectum within 48 hours of virus specimen collection during study visits
* No prior malignancy except nonmelanoma skin cancer
* No medical or psychiatric illness than would preclude study participation or compliance
* No other disorders requiring medical intervention that would preclude study participation
* No prior HPV vaccine
* More than 30 days since prior investigational vaccine
* More than 30 days since prior systemic steroid therapy
* No prior splenectomy
* More than 30 days since prior investigational drug
* More than 72 hours since prior antibiotic therapy for active infection

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 139 (Actual)
Dates: Start 2004-09; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
HPV-16 viral load | 6 months
  Following the univariate modeling, multivariate logistic regression models will be constructed by adding the demographic factors, baseline viral load, and type of cellular atypia to the model. The univariate logistic regression model for infection resolution is equivalent to a chi-square test.
Natural history of HPV 16 viral load | Baseline
  A repeated measures version of the zero-inflated log-normal model will be constructed.
Natural history of HPV 16 viral load | 3 months
  A repeated measures version of the zero-inflated log-normal model will be constructed.
Natural history of HPV 16 viral load | 6 months
  A repeated measures version of the zero-inflated log-normal model will be constructed.
Regression or non-regression of the cellular atypia | Up to 52 weeks
  The analysis for this will employ logistic regression models. A multivariate logistic regression model will be constructed. . A two group continuity corrected chi squared test with a 0.050 two-sided significance level will be used.

SECONDARY OUTCOMES:
HPV-16 viral load | 3 months
  Following the univariate modeling, multivariate logistic regression models will be constructed by adding the demographic factors, baseline viral load, and type of cellular atypia to the model. The univariate logistic regression model for infection resolution is equivalent to a chi-square test.
Time to infection resolution | Up to 52 weeks
  Kaplan Meier curves will be constructed.
Time to disease resolution | Up to 52 weeks
  Kaplan Meier curves will be constructed.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Meyskens, Principal Investigator — University of California Medical Center At Irvine-Orange Campus
Locations (1):
- University of California Medical Center At Irvine-Orange Campus, Orange, California, United States